CLINICAL TRIAL: NCT07208942
Title: Diagnosis Value of Interoceptive EEG Indicators by Rectal Stimulation in Patients With Disorders of Consciousness
Brief Title: Diagnosis Value of Interoceptive EEG Indicators by Rectal Stimulation in DoC
Status: Recruiting | Type: Observational
Sponsor: YiLin Zhao (Other)
Collaborators: The Second People's Hospital of Hefei (Unknown)
Responsible Party: Sponsor-Investigator, YiLin Zhao, PhD, Hangzhou Normal University
Organization: Hangzhou Normal University (Other)
Other Study IDs: 20241009-2
Record Dates: First submitted 2025-09-21; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Disorders of Consciousness
Keywords: Interoceptive; EEG; Rectal Stimulation; Diagnosis
MeSH Terms: conditions — Consciousness Disorders; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Disorders of consciousness: Patients assessed as Minimally Conscious State plus/minus (MCS+/-) and Unresponsive Wakefulness Syndrome (UWS) using the Coma Recovery Scale-Revised (CRS-R).
  Interventions: Device: Rectal Stimulation

INTERVENTIONS:
Device: Rectal Stimulation — The stimulation balloon was lubricated with paraffin oil and inserted until the distal end of the balloon was 10 cm from the anal verge, so as to eliminate the influence of different stimulation sites on the subjects.
  At the start of stimulation, the dilatable balloon was rapidly inflated to 60/80 mL, with a stimulation duration of 150 milliseconds. Concurrently with stimulation, the onset time of stimulation was marked on the electroencephalogram (EEG), and the time window for cortical potentials evoked by rapid rectal balloon distension stimulation was recorded. During the experiment, 35 stimulations were administered to the subjects; however, the first and last stimulations were excluded due to setup issues with the precision inflation-deflation control device for the intestinal balloon. Each stimulation was delivered as a 150-millisecond inflation pulse, providing 35 identical rectal stimulations. The inter-stimulus interval was randomly set to 12 ± 4 seconds, and EEG signals were

SUMMARY:
Study on the Significance and Value of Interoception-Related Indicators in the Classification of Patients with Disorders of Consciousness (DoC) via Rectal Stimulation

DETAILED DESCRIPTION:
Disorders of Consciousness (DoC) represent one of the sequelae of severe brain injuries caused by a variety of etiologies, including traumatic brain injury, stroke, and cardiac arrest. They may also result from primary neurological damage or systemic diseases. In recent years, with the advancement and development of surgical techniques and intensive care practices, an increasing number of DoC patients have survived life-threatening severe brain trauma. The large population of DoC patients imposes substantial psychological stress and economic burden on healthcare systems, social welfare services, and patients' families. Accurate identification and classification of DoC patients constitute a crucial prerequisite for clinical treatment and care.

Behavioral assessment of consciousness is currently the most common method for classifying DoC patients and is of great importance for critically ill patients. However, some cases of covert consciousness are difficult to identify, and even professional medical caregivers may encounter assessment errors. Such errors can lead to deviations in the selection of treatment strategies and the evaluation of prognostic efficacy for these patients. Precise diagnosis and classification of DoC are critical for prognostic treatment, as they enable the development of more rational rehabilitation protocols for patients and contribute to improving their quality of life.

The Coma Recovery Scale-Revised (CRS-R) is a standardized behavioral tool for the diagnosis of DoC. It primarily assesses patients' behavioral responses elicited by external sensory stimuli. The scale comprises six subscales: Auditory, Visual, Motor, Oromotor, Communication, and Arousal. Each subscale has a specific scoring range, with a total possible score of 23. Different total scores allow for the classification of patients into three categories: Vegetative State/Unresponsive Wakefulness Syndrome (VS/UWS), Minimally Conscious State (MCS, further divided into MCS+ and MCS-), and Emergent Minimally Conscious State (eMCS). However, the diagnosis and classification of VS/UWS and MCS using this scale are particularly challenging. This is because patients at the boundary between these two categories often exhibit highly similar behavioral responses to external stimuli, with only subtle differences. Additionally, the responses of DoC patients to behavioral assessments may be mere low-level reflexes or lack conscious involvement, making it difficult to achieve precise classification of DoC patients based solely on behavioral assessments.

Interoception refers to the bidirectional communication between the brain and the body's internal organs. Signals from internal organs-such as those related to heartbeat, respiratory movements, and gastrointestinal peristalsis-are transmitted to the cerebral cortex (including the insula and motor cortex) via the autonomic nervous system. Conversely, these cortical regions regulate the activity of target organs through the sympathetic and parasympathetic nervous systems. Interoception is essential for the maintenance of bodily homeostasis. Furthermore, a growing body of evidence indicates that interoception is also involved in higher cognitive functions, such as memory formation, emotional processing, and even the construction of the sense of self. Compared with exteroceptive pathways, the ascending interoceptive pathways in DoC patients tend to remain relatively intact. Therefore, interoception-related indicators, as a complement to exteroceptive behavioral response indicators, hold significant clinical value for the precise assessment of DoC patients.

Research on interoception-related indicators has emerged as a novel field for the differential diagnosis of DoC patients. These indicators serve as a vital supplement to behavioral and imaging assessments. Moreover, their application requires patients to engage in active conscious participation and induce awareness, which means interoception-related indicators can undertake the assessment tasks typically performed by imaging techniques in a more cost-effective and convenient manner. Consequently, they have inevitably become a focus of research in the field of consciousness and consciousness assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-acute Disorders of Consciousness (DoC) (disease course ≥ 28 days).
* Aged 18 years or older.
* No symptoms of fever, infection, or other similar conditions within 15 days.
* No use of sedatives within 15 days.
* No use of any drugs that may alter gastrointestinal motility within 7 days prior to testing.
* Family members of participating patients have provided consent and signed the informed consent form.

Exclusion Criteria:

* Patients with functional impairments caused by developmental psychiatric disorders or neurological diseases.
* Patients with untreated epilepsy.
* Untreated cerebral edema.
* Patients with unstable vital signs.
* A history of intestinal diseases.
* A history of abdominal surgery other than simple appendectomy or simple cholecystectomy.
* Organic diseases such as spinal cord injury, traumatic brain injury, and thyroid dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients assessed as Minimally Conscious State plus/minus (MCS+/-) and Unresponsive Wakefulness Syndrome (UWS) using the Coma Recovery Scale-Revised (CRS-R)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosis Value of Interoceptive EEG Indicators by Rectal Stimulation inDoC | December 2024 - December 2025
  This study aims to develop and validate an objective neurophysiological biomarker for classifying consciousness levels in patients with Disorders of Consciousness (DoC), such as the Unresponsive Wakefulness Syndrome (UWS) and the Minimally Conscious State (MCS). The primary objective is to determine whether cortical responses to a rectal balloon distension stimulus, which engages preserved interoceptive neural pathways, can effectively differentiate between these patient groups and healthy controls. In this prospective, case-control study, participants (DoC patients and healthy controls) will undergo electroencephalography (EEG) recording during a standardized rectal stimulation paradigm. The primary outcome measures will include the amplitude of event-related potential (ERP) components (N1, P2, P3) at central (Cz) and frontal (Fz) electrodes, and the spectral power in the theta band (3-5 Hz) derived from Event-Related Spectral Perturbation (ERSP) analysis. The findings are expected t

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - Hangzhou Normal University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No